CLINICAL TRIAL: NCT02447991
Title: A Phase II/III Trial on Rizatriptan for Vestibular Migraine
Brief Title: Rizatriptan for Episodic Dizziness in Vestibular Migraine
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Robert W. Baloh (Other)
Responsible Party: Sponsor-Investigator, Robert W. Baloh, Robert W. Baloh, M.D., UCLA Principal Investigator/Study Chair, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB12-001549
Record Dates: First submitted 2015-03-18; First posted 2015-05-19 (Estimated); Results first posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2019-10

CONDITIONS: Vestibular Migraine; Migrainous Vertigo
MeSH Terms: interventions — rizatriptan; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): During the Treatment Phase, three placebo capsules will be administered to each subject. One capsule will be taken during one acute episode, until three episodes are treated with the study drug.
  Interventions: Drug: Placebo
- Rizatriptan (Experimental): During the Treatment Phase, three Rizatriptan capsules will be administered to each subject. One capsule will be taken during one acute episode, until three episodes are treated with the study drug.
  Interventions: Drug: Rizatriptan

INTERVENTIONS:
Drug: Rizatriptan — During the study either placebo or Rizatriptan will be given to subjects to take during the treatment phase of this study.
  Other Names: Maxalt
  Arms: Rizatriptan
Drug: Placebo — During the study either placebo or Rizatriptan will be given to subjects to take during the treatment phase of the study.
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
Suffering from dizzy spells and migraine headaches?

Vestibular Migraine (VM), a newly recognized type of migraine that causes bouts of dizziness.

University of California, Los Angeles (UCLA) and The Mayo Clinic is seeking people with VM to participate in a research study. The purpose of this study is to look at the natural history of VM and learn more about common symptoms. Investigators also want to learn the effects, both positive and negative, of the commonly used migraine drug, rizatriptan, when it is used for spells of dizziness in people with VM.

Patients may be eligible to participate if:

* Patients are between the ages of 18 & 65
* Patients have a history of vestibular migraine
* Patients are able to maintain a vestibular symptom diary

The study includes 3 visits with compensation. All participants must complete questionnaires on dizziness, headache symptoms, general health and well-being, mental health, and a questionnaire on patient's satisfaction with study medication.

DETAILED DESCRIPTION:
The primary Specific Aim is to conduct the first successful controlled study of a treatment for Vestibular Migraine. The investigators hypothesize that rizatriptan will be superior to a look alike inactive capsule for:

1a. Reducing the severity and duration of vertigo attacks in patients with Vestibular Migraine,

1b. Reducing the severity of symptoms commonly associated with vertigo attacks in patients with Vestibular Migraine (e.g., nausea, vomiting, motion sensitivity, gait disturbance, headache, light and sound sensitivity), and

1c. Improving treatment satisfaction and health-related quality of life in patients with Vestibular Migraine, and that

1d. Rizatriptan will be well tolerated by patients with Vestibular Migraine.

ELIGIBILITY:
Inclusion Criteria: Must answer yes to be eligible

1. Are between the ages of 18 & 65
2. Have a history of vestibular migraine
3. Are able to maintain a vestibular symptom diary

   History that fulfills all criteria for VM as defined in Table 1, except that attacks must last at least 2 hours.
4. At least 5 episodes
5. A current or past history of migraine without aura or migraine with aura
6. Vestibular symptoms of moderate or severe intensity lasting at least 2 hours
7. 50% of episodes are associated with at least one of the following:

   Headache with at least 2 of:
   * unilateral location
   * pulsating quality
   * moderate or severe intensity,
   * aggravation by routine physical activity
8. Experience photophobia and phonophobia
9. Experience visual aura
10. Episodes must have a spontaneous onset and resolution without associated hearing loss or interictal neurotologic deficits.
11. Other causes of vestibular symptoms ruled out by appropriate clinical investigations.
12. Current medication list compatible with Concomitant Medications below.
13. Able to maintain a Vestibular Symptom Diary and complete all other study procedures.

Exclusion Criteria: Must answer no to be eligible.

1. Ménière's disease by The American Academy of Otolaryngology-Head and Neck Surgery Foundation (AAO-HNS) criteria60.
2. Migraine with brainstem aura (formerly basilar-type migraine) by the International Classification of Headache Disorders (ICHD-3) criteria.14
3. Ischemic heart disease, coronary artery vasospasm, uncontrolled hypertension.
4. History of stroke or transient ischemic attack.
5. History of using rizatriptan specifically to treat vestibular attacks.
6. History of adverse response to triptans or intolerance to lactose.
7. Women who are pregnant or breastfeeding.
8. Unable or unwilling to comply with study requirements for any reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Baloh, M.D., Principal Investigator — University of California, Los Angeles
Locations (3):
- United States (3):
  - University of California, Los Angeles, Los Angeles, California
  - Mayo Clinic, Rochester, Minnesota
  - ICAHN School of Medicine at Mount Sinai, New York, New York

REFERENCES:
- [Derived] Staab JP, Eggers SDZ, Jen JC, LeMahieu AM, Geske JR, Liu H, Hofschulte DR, Gonzalez GR, Neff BA, Shepard NT, McCaslin DL, Baloh RW. Rizatriptan vs Placebo for Attacks of Vestibular Migraine: A Randomized Clinical Trial. JAMA Neurol. 2025 Jul 1;82(7):676-686. doi: 10.1001/jamaneurol.2025.1006. PMID 40354049

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 222 enrolled, 134 completed the observation period and moved on to the treatment phase, having had 2 qualifying episodes in the observation phase. Participants who did not have 2 qualifying episodes in the 12 month observation phase were withdrawn from the study.
Period: Overall Study
Arm/Group | Placebo | Rizatriptan
Started | 45 | 89
Completed | 35 | 59
Not Completed | 10 | 30
Not completed — Withdrawn by subject - no data | 0 | 2
Not completed — Withdrawn by Subject - with data | 4 | 4
Not completed — Lost to Follow-up - no data | 3 | 6
Not completed — Lost to follow-up - with data | 0 | 3
Not completed — End of study - no treatment results | 3 | 6
Not completed — End of study - partial treatment results | 0 | 9

BASELINE CHARACTERISTICS:
Groups:
- Placebo: During the Treatment Phase, three placebo capsules were administered to each subject, one capsule to be taken during one acute episode, until three episodes are treated with the study drug.
- Rizatriptan: During the Treatment Phase, three Rizatriptan capsules were administered to each subject, one capsule to be taken during one acute episode, until three episodes are treated with the study drug.
- Total: Total of all reporting groups
Arm/Group | Placebo | Rizatriptan | Total
Number analyzed (Participants) | 45 | 89 | 134
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 89 | 134
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 69 | 101
  Male | 13 | 20 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 9 | 11
  Not Hispanic or Latino | 3 | 0 | 3
  Unknown or Not Reported | 40 | 80 | 120
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 9 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 7 | 7
  White | 39 | 69 | 108
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 45 | 89 | 134

OUTCOME MEASURES:

1. Primary Outcome: Episodes With Vertigo Symptom Reduced From Moderate/Severe to None/Mild
Description: Episodes in which a reduction in symptom severity from moderate/severe (rating 2/3) at time of taking study medication to none/mild rating (0/1) was achieved. After taking study medication participants reported symptoms using a patient self-report of the severity of vestibular symptoms (vertigo and unsteadiness/dizziness) wherein 0=no symptoms, 1=mild symptoms (no interference with activities), 2=moderate symptoms (had to alter some activities), and 3=severe symptoms (had to stop most or all activities).
Time Frame: 1 hour after taking study medication
Population: Participants who experienced episodes with moderate/severe symptoms were included in the analyses
Measure: Number; unit: Episodes
Units Other Than Participants: Episodes of vertigo
Groups:
- Placebo: Participants were instructed to treat three separate episodes of moderate to server vestibular symptoms with study drug, (placebo capsule) orally.
- Rizatriptan: Participants were instructed to treat three separate episodes of moderate to server vestibular symptoms with study drug, (rizatriptan 10 mg) orally.
Arm/Group | Placebo | Rizatriptan
Number analyzed (Participants) | 39 | 75
Number analyzed (Episodes of vertigo) | 88 | 151
Episodes | 50 | 73
Statistical Analysis 1: Comparison: Placebo vs Rizatriptan; Hypothesis: Rizatriptan will be superior to placebo in reducing the severity of vertigo as measured by the proportion of treated episodes in which subjects experience a reduction in severity rating from Grade 3/2 to Grade 1/0 at 1 hour after taking study medication; Test type: Superiority; p < 0.33, Chi-squared, Corrected — Significance level p < 0.05; This analysis applies to proportion of treated episodes

2. Primary Outcome: Episodes With Symptoms of Unsteadiness/Dizziness Reduced From Moderate/Severe to None/Mild
Description: Episodes of unsteadiness/dizziness in which a reduction in symptom severity from moderate/severe (rating 2/3) to none/mild rating (0/1) was achieved. After taking study medication participants reported symptoms using a patient self-report of the severity of vestibular symptoms (vertigo and unsteadiness/dizziness) wherein 0=no symptoms, 1=mild symptoms (no interference with activities), 2=moderate symptoms (had to alter some activities), and 3=severe symptoms (had to stop most or all activities).
Time Frame: 1 hour after taking study medication
Population: Participants who experienced episodes with moderate/severe symptoms were included in the analyses
Measure: Number; unit: Episodes
Units Other Than Participants: Episodes of Unsteadiness/Dizziness
Arm/Group | Placebo | Rizatriptan
Number analyzed (Participants) | 39 | 75
Number analyzed (Episodes of Unsteadiness/Dizziness) | 89 | 151
Episodes | 11 | 29
Statistical Analysis 1: Comparison: Placebo vs Rizatriptan; Hypothesis: Rizatriptan will be superior to placebo in reducing the severity of unsteadiness/dizziness as measured by the proportion of treated episodes in which subjects experience a reduction in severity rating from Grade 3/2 to Grade 1/0 at 1 hour after taking study medication; Test type: Superiority; p < 0.18, Chi-squared, Corrected — Signficant at p < 0.05; This analysis applies to proportion of treated episodes

3. Secondary Outcome: Episodes With Complete Relief of Vertigo as Vestibular Symptom
Description: The number of episodes in which complete relief of vertigo symptoms (rating 0) was achieved. After taking study medication participants reported symptoms using a patient self-report of the severity of vestibular symptoms (vertigo and unsteadiness/dizziness) wherein 0=no symptoms, 1=mild symptoms (no interference with activities), 2=moderate symptoms (had to alter some activities), and 3=severe symptoms (had to stop most or all activities).
Time Frame: 1 hour after taking study medication
Population: Participants who experienced episodes with moderate/severe symptoms were included in the analyses.
Measure: Number; unit: Episodes
Units Other Than Participants: Episodes of vertigo
Groups:
- Placebo: Participants were instructed to treat three separate attacks of moderate to server vestibular symptoms with study drug, (placebo capsule) orally.
- Rizatriptan: Participants were instructed to treat three separate attacks of moderate to server vestibular symptoms with study drug, (rizatriptan 10 mg) orally.
Arm/Group | Placebo | Rizatriptan
Number analyzed (Participants) | 39 | 75
Number analyzed (Episodes of vertigo) | 88 | 151
Episodes | 35 | 56
Statistical Analysis 1: Comparison: Placebo vs Rizatriptan; Hypothesis: Rizatriptan will be superior to placebo in reducing the severity of vertigo as measured by the proportion of treated episodes in which subjects experience freedom from vestibular symptoms (i.e., severity rating of Grade 0) at 1 hour after taking study medication; Test type: Superiority; p < 0.62, Chi-squared, Corrected — Significance threshold p<0.05; This analysis applies to proportion of treated episodes

4. Secondary Outcome: Episodes With Complete Relief of Unsteadiness/Dizziness Vestibular Symptoms
Description: The outcome was the number of episodes in which complete relief of symptoms of unsteadiness/dizziness (rating 0) was achieved. After taking study medication participants reported symptoms using a patient self-report of the severity of vestibular symptoms (vertigo and unsteadiness/dizziness) wherein 0=no symptoms, 1=mild symptoms (no interference with activities), 2=moderate symptoms (had to alter some activities), and 3=severe symptoms (had to stop most or all activities).
Time Frame: 1 hour after taking study medication
Population: Participants who experienced episodes with moderate/severe symptoms were included in the analyses.
Measure: Number; unit: Episodes
Units Other Than Participants: Episodes of Unsteadiness/Dizziness
Arm/Group | Placebo | Rizatriptan
Number analyzed (Participants) | 39 | 75
Number analyzed (Episodes of Unsteadiness/Dizziness) | 89 | 151
Episodes | 2 | 12
Statistical Analysis 1: Comparison: Placebo vs Rizatriptan; Hypothesis: Rizatriptan will be superior to placebo in reducing the severity of unsteadiness/dizziness as measured by the proportion of treated episodes in which subjects experience freedom from vestibular symptoms (i.e., severity rating of Grade 0) at 1 hour after taking study medication; Test type: Superiority; p < 0.19, Chi-squared, Corrected — Significance threshold p < 0.05; This analysis applies to proportions of treated episodes

5. Secondary Outcome: Episodes With Headache Reduced From Moderate/Severe to None/Mild
Description: The outcome was the number of episodes in which a reduction of headache symptoms (rating 0) was achieved. After taking study medication participants reported symptoms using a patient self-report of the severity of vestibular symptoms wherein 0=no symptoms, 1=mild symptoms (no interference with activities), 2=moderate symptoms (had to alter some activities), and 3=severe symptoms (had to stop most or all activities).
Time Frame: 1 hour after taking study medication
Population: Participants who experienced episodes with moderate/severe symptoms were included in the analyses.
Measure: Number; unit: Episodes
Units Other Than Participants: Episodes of headache
Arm/Group | Placebo | Rizatriptan
Number analyzed (Participants) | 39 | 75
Number analyzed (Episodes of headache) | 89 | 149
Episodes | 38 | 44
Statistical Analysis 1: Comparison: Placebo vs Rizatriptan; Hypothesis: Rizatriptan will be superior to placebo in reducing the severity of headaches as measured by the proportion of treated episodes in which subjects experience a reduction in severity rating from Grade 3/2 to Grade 1/0 at 1 hour after taking study medication; Test type: Superiority; p < 0.14, Chi-squared, Corrected — Significance threshold p<0.05; This analysis applies to proportion of treated episodes

6. Secondary Outcome: Episodes With Photophobia/Phonophobia Reduced From Moderate/Severe to None/Mild
Description: The outcome was the number of episodes in which a reduction of symptoms (rating 0/1) was achieved. After taking study medication participants reported symptoms using a patient self-report of the severity of vestibular symptoms wherein 0=no symptoms, 1=mild symptoms (no interference with activities), 2=moderate symptoms (had to alter some activities), and 3=severe symptoms (had to stop most or all activities).
Time Frame: 1 hour after taking study medication
Population: Participants who experienced episodes with moderate/severe symptoms were included in the analyses.
Measure: Number; unit: Episodes
Units Other Than Participants: Episodes of Photophobia/Phonophobia
Arm/Group | Placebo | Rizatriptan
Number analyzed (Participants) | 39 | 75
Number analyzed (Episodes of Photophobia/Phonophobia) | 89 | 151
Episodes | 33 | 59
Statistical Analysis 1: Comparison: Placebo vs Rizatriptan; Hypothesis: Rizatriptan will be superior to placebo in reducing the severity of photophobia/phonophobia as measured by the proportion of treated episodes in which subjects experience a reduction in severity rating from Grade 3/2 to Grade 1/0 at 1 hour after taking study medication; Test type: Superiority; p < 0.72, Chi-squared, Corrected — Significance threshold p < 0.05; This analysis applies to proportion of treated episodes

7. Secondary Outcome: Episodes With Sensitivity to Motion Reduced From Moderate/Severe to None/Mild
Description: The outcome was the number of episodes in which a reduction of sensitivity to motion symptoms (rating 0/1) was achieved. After taking study medication participants reported symptoms using a patient self-report of the severity of vestibular symptoms wherein 0=no symptoms, 1=mild symptoms (no interference with activities), 2=moderate symptoms (had to alter some activities), and 3=severe symptoms (had to stop most or all activities).
Time Frame: 1 hour after taking study medication
Population: Participants who experienced episodes with moderate/severe symptoms were included in the analyses.
Measure: Number; unit: Episodes
Units Other Than Participants: Episodes of Sensitivity to Motion
Arm/Group | Placebo | Rizatriptan
Number analyzed (Participants) | 39 | 75
Number analyzed (Episodes of Sensitivity to Motion) | 89 | 151
Episodes | 19 | 39
Statistical Analysis 1: Comparison: Placebo vs Rizatriptan; Hypothesis: Rizatriptan will be superior to placebo in reducing the severity of sensitivity to motion as measured by the proportion of treated episodes in which subjects experience a reduction in severity rating from Grade 3/2 to Grade 1/0 at 1 hour after taking study medication; Test type: Superiority; p < 0.48, Chi-squared, Corrected — Significance threshold p < 0.05; This analysis applies to proportion of treated episodes

8. Secondary Outcome: Episodes With Nausea/Vomiting Reduced From Moderate/Severe to None/Mild
Description: as for outcome 6
Time Frame: 1 hour after taking study medication
Population: Participants who experienced episodes with moderate/severe symptoms were included in the analyses.
Measure: Number; unit: Episodes
Units Other Than Participants: Episodes of Nausea/Vomiting
Arm/Group | Placebo | Rizatriptan
Number analyzed (Participants) | 39 | 75
Number analyzed (Episodes of Nausea/Vomiting) | 89 | 150
Episodes | 50 | 67
Statistical Analysis 1: Comparison: Placebo vs Rizatriptan; Hypothesis: Rizatriptan will be superior to placebo in reducing the severity of nausea/vomiting as measured by the proportion of treated episodes in which subjects experience a reduction in severity rating from Grade 3/2 to Grade 1/0 at 1 hour after taking study medication; Test type: Superiority; p < 0.35, Chi-squared, Corrected — Significance threshold p < 0.05; This analysis applies to proportion of treated episodes

9. Secondary Outcome: Satisfaction With Treatment
Description: Treatment Satisfaction Questionnaire for Medication (TSQM) assessed four domains of participants' satisfaction with treatment, with scale ranges from 0 (extremely dissatisfied) to 100 (not at all dissatisfied) for each of the categories (Effectiveness, Side Effects, Convenience, and Overall Satisfaction).
Time Frame: 48 hour after taking study medication
Population: Participants who experienced episodes with moderate/severe vestibular symptoms were included in the analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: Participants meeting International Headache Society and International Classification of Vestibular Disorders criteria for vestibular migraine and experiencing at least two attacks documented during the 12-month prospective observation phase of this study were randomized in a 2:1 ratio to rizatriptan versus placebo. Participants were instructed to treat three separate attacks of moderate to server vestibular symptoms with study drug, (placebo capsule) orally.
- Rizatriptan: Participants meeting International Headache Society and International Classification of Vestibular Disorders criteria for vestibular migraine and experiencing at least two attacks documented during the 12-month prospective observation phase of this study were randomized in a 2:1 ratio to rizatriptan versus placebo. Participants were instructed to treat three separate attacks of moderate to server vestibular symptoms with study drug, (rizatriptan 10 mg) orally.
Arm/Group | Placebo | Rizatriptan
Number analyzed (Participants) | 39 | 75
score on a scale
  Effectiveness | 37.2 (27.0) | 49.7 (28.6)
  Side Effects | 78.8 (26.0) | 81.6 (22.6)
  Convenience | 70.0 (17.4) | 71.0 (17.8)
  Overall Satisfaction | 45.9 (27.1) | 58.2 (26.7)
Statistical Analysis 1: Comparison: Placebo vs Rizatriptan; Hypothesis: Rizatriptan will be superior to placebo on the Treatment Satisfaction Questionnaire for Medication at 48 hours after each attack treated with effectiveness of study medication; Test type: Superiority; p < 0.022, Regression, Linear — Significance of threshold p<0.05; This analysis applies to proportion of treated episodes
Statistical Analysis 2: Comparison: Placebo vs Rizatriptan; Hypothesis: Rizatriptan will be superior to placebo on the Treatment Satisfaction Questionnaire for Medication at 48 hours after each attack treated with side effects of study medication; Test type: Superiority; p < 0.418, Regression, Linear — Significance of threshold p<0.05; This analysis applies to proportion of treated episodes
Statistical Analysis 3: Comparison: Placebo vs Rizatriptan; Hypothesis: Rizatriptan will be superior to placebo on the Treatment Satisfaction Questionnaire for Medication at 48 hours after each attack treated with convenience of study medication; Test type: Superiority; p < 0.674, Regression, Linear — Significance of threshold p<0.05; This analysis applies to proportion of treated episodes
Statistical Analysis 4: Comparison: Placebo vs Rizatriptan; Hypothesis: Rizatriptan will be superior to placebo on the Treatment Satisfaction Questionnaire for Medication at 48 hours after each attack treated with overall satisfaction of study medication; Test type: Superiority; p < 0.016, Regression, Linear — Significance of threshold of p<0.05; This analysis applies to proportion of treated episodes

10. Secondary Outcome: Health-Related Quality of Life
Description: Short Form Survey - 12 (SF-12) assessed physical and mental well-being after taking study medication for each episode, generating composite scores in each domain from 12 questions. The range is 0-100 with higher scores indicated better physical and mental health functioning.
Time Frame: 48 hour after taking study medication
Population: Episodes with moderate/severe symptoms were included in the analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: episodes of vestibular symptoms
Arm/Group | Placebo | Rizatriptan
Number analyzed (Participants) | 39 | 75
Number analyzed (episodes of vestibular symptoms) | 89 | 151
score on a scale
  Physical well-being after study medication | 37.5 (10.5) | 41.9 (8.9)
  Mental well-being after study medication | 44.2 (13.9) | 45.4 (11.4)
Statistical Analysis 1: Comparison: Placebo vs Rizatriptan; Hypothesis: Rizatriptan will be superior to placebo on physical well-being; Test type: Superiority; p < 0.009, Regression, Linear — Significance threshold p<0.05; This analysis applies to proportion of treated episodes
Statistical Analysis 2: Comparison: Placebo vs Rizatriptan; Hypothesis: Rizatriptan will be superior to placebo on mental well-being; Test type: Superiority; p < 0.467, Regression, Linear — Significance threshold p<0.05; This analysis applies to proportion of treated episodes

11. Secondary Outcome: Side Effects
Description: Number of adverse events experienced by participants. Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 categorizes all domains of physical and psychological side effects, grading them 1-mild, 2-moderate, 3-severe, 4-life threatening, 5-death.
Time Frame: 48 hour after taking study medication
Population: Participants who experienced episodes with moderate/severe vestibular symptoms were included in the analyses.
Measure: Number; unit: Adverse Events
Arm/Group | Placebo | Rizatriptan
Number analyzed (Participants) | 39 | 75
Adverse Events
  Fatigue | 7 | 44
  Sleepiness/Drowsiness | 11 | 51
  Upset Stomach, nausea, vomiting | 8 | 19
  Constipation or diarrhea | 3 | 3
  Hearth rhythm problems | 2 | 5
  Chest pain or decreased exercise tolerance | 1 | 0
  Swelling or puffiness | 0 | 3
  Fever or chills | 0 | 4
  Worsening of dizziness or gait | 3 | 15
  Worsening of headache | 9 | 13
  Ataxia | 1 | 4
  Speech problems | 1 | 3
  Weakness of arms/legs/face or loss of sensation | 5 | 7
  Agitation | 1 | 5
  Anxiety | 5 | 12
  Serious adverse effects | 0 | 0
  Discontinuation due to adverse effects | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs Rizatriptan; Hypothesis: Rizatriptan will be tolerated as well as placebo with regard to fatigue; Test type: Superiority; p < 0.013, Logistic regression with GEE — Significance threshold p<0.05; GEE=generalized estimating equations - this accounts for repeated measures within patients.This analysis applies to proportion of treated episodes
Statistical Analysis 2: Comparison: Placebo vs Rizatriptan; Hypothesis: Rizatriptan will be tolerated as well as placebo with regard to sleepiness/drowsiness; Test type: Superiority; p < 0.021, Logistic regression with GEE — Significance threshold p<0.05; GEE=generalized estimating equations - this accounts for repeated measures within patients. This analysis applies to proportion of treated episodes

12. Secondary Outcome: Episodes With Sustained Reduction in Severity of Vertigo From Moderate/Severe to None/Mild Without Additional Medication
Description: Episodes in which participants achieved reduction of symptoms (from rating 2-3 to 0-1). After taking study medication participants reported symptoms using a patient self-report of the severity of vestibular symptoms wherein 0=no symptoms, 1=mild symptoms (no interference with activities), 2=moderate symptoms (had to alter some activities), and 3=severe symptoms (had to stop most or all activities).
Time Frame: 24 hours after taking study medication
Population: Participants who experienced episodes with moderate/severe symptoms were included in the analyses.
Measure: Number; unit: Episodes
Units Other Than Participants: Episodes of vertigo
Arm/Group | Placebo | Rizatriptan
Number analyzed (Participants) | 39 | 75
Number analyzed (Episodes of vertigo) | 61 | 109
Episodes | 54 | 97
Statistical Analysis 1: Comparison: Placebo vs Rizatriptan; Hypothesis: Rizatriptan will be superior to placebo in reducing the severity of vertigo measured by the proportion of treated episodes that subjects rate at grade 1/0 24 hours after taking study medication; Test type: Superiority; p < 0.76, Chi-squared, Corrected — Significance threshold p<0.05; This analysis applies to proportion of treated episodes

13. Secondary Outcome: Episodes With Sustained Reduction in Severity of Dizziness/Unsteadiness From Moderate/Severe to None/Mild Without Additional Medication
Description: as for outcome 12
Time Frame: 24 hours after taking study medication
Population: Participants who experienced episodes with moderate/severe vestibular symptoms were included in the analyses.
Measure: Number; unit: Episodes
Units Other Than Participants: Episodes of Unsteadiness/Dizziness
Arm/Group | Placebo | Rizatriptan
Number analyzed (Participants) | 39 | 75
Number analyzed (Episodes of Unsteadiness/Dizziness) | 62 | 109
Episodes | 41 | 90
Statistical Analysis 1: Comparison: Placebo vs Rizatriptan; Hypothesis: Rizatriptan will be superior to placebo in reducing the severity of unsteadiness/dizziness episodes measured by the proportion of treated episodes that subjects rate at grade 1/0 24 hours after taking study medication; Test type: Superiority; p < 0.041, Chi-squared, Corrected — Significance threshold p < 0.05; This analysis applies to proportion of treated episodes

14. Secondary Outcome: Episodes With Headache Symptoms Reduced From Moderate/Severe (3/4) to None/Mild (0/1) Without Additional Medication
Description: After taking study medication participants reported symptoms using a patient self-report of the severity of vestibular symptoms wherein 0=no symptoms, 1=mild symptoms (no interference with activities), 2=moderate symptoms (had to alter some activities), and 3=severe symptoms (had to stop most or all activities).
Time Frame: 24 hours after taking study medication
Population: Participants who experienced episodes with moderate/severe vestibular symptoms were included in the analyses.
Measure: Number; unit: Episodes
Units Other Than Participants: Episodes of headache
Arm/Group | Placebo | Rizatriptan
Number analyzed (Participants) | 39 | 75
Number analyzed (Episodes of headache) | 62 | 109
Episodes | 46 | 94
Statistical Analysis 1: Comparison: Placebo vs Rizatriptan; Hypothesis: Rizatriptan will be superior to placebo in reducing the severity of headaches measured by the proportion of treated episodes that subjects rate at grade 1/0 24 hours after taking study medication; Test type: Superiority; p < 0.12, Chi-squared, Corrected — Significance threshold p<0.05; This analysis applies to proportion of treated episodes

15. Secondary Outcome: Episodes With Photophobia/Phonophobia Symptoms Reduced From Moderate/Severe (3/4) to None/Mild (0/1) Without Additional Medication
Description: as for outcome 14
Time Frame: 24 hours after taking study medication
Population: Participants who experienced episodes with moderate/severe vestibular symptoms were included in the analyses.
Measure: Number; unit: Episodes
Units Other Than Participants: Episodes of photophobia/phonophobia
Arm/Group | Placebo | Rizatriptan
Number analyzed (Participants) | 39 | 75
Number analyzed (Episodes of photophobia/phonophobia) | 62 | 109
Episodes | 45 | 95
Statistical Analysis 1: Comparison: Placebo vs Rizatriptan; Hypothesis: Rizatriptan will be superior to placebo in reducing the severity of photophobia/phonophobia measured by the proportion of treated episodes that subjects rate at grade 1/0 24 hours after taking study medication; Test type: Superiority; p < 0.051, Chi-squared, Corrected — Significance threshold p<0.05; This analysis applies to proportion of treated episodes

16. Secondary Outcome: Episodes With Sensitivity to Motion Symptoms Reduced From Moderate/Severe (3/4) to None/Mild (0/1) Without Additional Medication
Description: as for outcome 14
Time Frame: 24 hours after taking study medication
Population: Participants who experienced episodes with moderate/severe symptoms were included in the analyses.
Measure: Number; unit: Episodes
Units Other Than Participants: Episodes of sensitivity to motion
Arm/Group | Placebo | Rizatriptan
Number analyzed (Participants) | 39 | 75
Number analyzed (Episodes of sensitivity to motion) | 62 | 109
Episodes | 42 | 95
Statistical Analysis 1: Comparison: Placebo vs Rizatriptan; Hypothesis: Rizatriptan will be superior to placebo in reducing the severity of sensitivity to motion measured by the proportion of treated episodes that subjects rate at grade 1/0 24 hours after taking study medication; Test type: Superiority; p < 0.006, Chi-squared, Corrected — Significance threshold p<0.05; This analysis applies to proportion of treated episodes

17. Secondary Outcome: Episodes With Nausea/Vomiting Symptoms Reduced From Moderate/Severe (3/4) to None/Mild (0/1) Without Additional Medication
Description: as for outcome 14
Time Frame: 24 hours after taking study medication
Population: Participants who experienced episodes with moderate/severe symptoms were included in the analyses.
Measure: Number; unit: Episodes
Units Other Than Participants: Episodes of nausea/vomiting
Arm/Group | Placebo | Rizatriptan
Number analyzed (Participants) | 39 | 75
Number analyzed (Episodes of nausea/vomiting) | 62 | 108
Episodes | 57 | 101
Statistical Analysis 1: Comparison: Placebo vs Rizatriptan; Hypothesis: Rizatriptan will be superior to placebo in reducing the severity of nausea/vomiting measured by the proportion of treated episodes that subjects rate at grade 1/0 24 hours after taking study medication; Test type: Superiority; p < 0.67, Chi-squared, Corrected — Significance threshold p<0.05; This analysis applies to proportion of treated episodes

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: 48 hours after each episode, until 3 episodes occur, up to 5 years of study duration
Arm/Group | Placebo | Rizatriptan
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/89
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/89
Other Adverse Events (participants affected / at risk) | 45/45 | 89/89
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=45) | Rizatriptan (N=89)
Fatigue (General disorders) | 7 (7) | 44 (44)
Sleepiness/drowsiness (General disorders) | 11 (11) | 51 (51)
Upset stomach, nausea, vomiting (Gastrointestinal disorders) | 8 (8) | 19 (19)
Constipation or diarrhea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Hearth rhythm problems (Cardiac disorders) | 2 (2) | 5 (5)
Chest pain or decreased exercise tolerance (Cardiac disorders) | 1 (1) | 0 (0)
Swelling or puffiness (General disorders) | 0 (0) | 3 (3)
Fever or chills (General disorders) | 0 (0) | 4 (4)
Worsening of dizziness or gait (Nervous system disorders) | 3 (3) | 15 (15)
Worsening of headache (Nervous system disorders) | 9 (9) | 13 (13)
Ataxia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Speech problems (Nervous system disorders) | 1 (1) | 3 (3)
Weakness of arm/legs/face or loss of sensation (Musculoskeletal and connective tissue disorders) | 5 (5) | 7 (7)
Agitations (Psychiatric disorders) | 1 (1) | 5 (5)
Anxiety (Psychiatric disorders) | 5 (5) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/91/NCT02447991/Prot_SAP_000.pdf